CLINICAL TRIAL: NCT01702831
Title: A Phase II Study of Busulfan & Melphalan as Conditioning Regimen for ASCT in Patients Who Received Bortezomib Based Induction for Newly Diagnosed Multiple Myeloma Followed by Lenalidomide Maintenance Until Progression.
Brief Title: Busulfan & Melphalan Conditioning for Autologous Stem Cell Transplant (ASCT) and Lenalidomide Maintenance
Acronym: BuMelMCRN001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other); Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCRN 001
Record Dates: First submitted 2012-08-29; First posted 2012-10-08 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Multiple Myeloma
Keywords: Newly Diagnosed multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Busulfan; Melphalan; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BuMel + lenalidomide Maintenance (Experimental): I.V. Busulfan + I.V. Melphalan for conditioning prior ASCT, followed by Lenalidomide maintenance at day 100 after ASCT.
  Interventions: Drug: Busulfan; Drug: Melphalan; Drug: Lenalidomide

INTERVENTIONS:
Drug: Busulfan — Once daily intravenous (IV) busulfan at a dose of 3.2 mg/kg or equivalent pharmacokinetics directed dose for three consecutive days (days -5 to -3), option 1 OR Once daily intravenous (IV) busulfan at a dose of 3.2mg/kg or equivalent pharmacokinetics directed dose for three consecutive days (days -6 to -4), option 2.
  Other Names: Busulfex
Drug: Melphalan — I.V. reduced dose of melphalan (140mg/m2) on day -2, followed by an autologous stem cell transplant on day 0 (day -1 will be a rest day) - this is referred to as "Option 1" dosing schema OR I.V. reduced dose of melphalan (140mg/m2) on day -3 followed by autologous stem cell transplant on day 0 (days -2 and -1 will be rest days). This is referred to as "Option 2"
  Other Names: Alkeran
Drug: Lenalidomide — Oral lenalidomide 10mg per day (on all 28 days of a 28 day cycle) for the first three cycles and then escalated to 15 mg daily if clinically appropriate to do so. The lenalidomide maintenance will start on day 100 post ASCT and continue till disease progression.
  Other Names: Revlimid

SUMMARY:
A number of strategies have been proposed to improve the outcome of ASCT. The three main strategies are to incorporate novel agents into the induction regimen, using maintenance therapy following ASCT and the final strategy is to enhance conditioning regimens.

Investigators would like to explore all these three strategies in this study: Investigators propose to take patients who have had standard novel agent (bortezomib) based induction regimens into this study and then use a dose-adjusted combination of busulfan and melphalan as conditioning regimen and finally Investigators would like to incorporate lenalidomide maintenance post ASCT until disease progression.

DETAILED DESCRIPTION:
STUDY RATIONALE AND PURPOSE:

A number of strategies have been proposed to improve the outcome of ASCT. The three main strategies are to incorporate novel agents into the induction regimen, using maintenance therapy following ASCT and the final strategy is to enhance conditioning regimens.

Investigators would like to explore all these three strategies in this study: Investigators propose to take patients who have had standard novel agent (bortezomib) based induction regimens into this study and then use a dose-adjusted combination of busulfan and melphalan as conditioning regimen and finally Investigators would like to incorporate lenalidomide maintenance post ASCT until disease progression.

The conventional immunological markers used to define myeloma disease status have also been a subject of debate recently with some reports suggesting that more accurate disease assessment tools are needed to better decide on management of this disease. One of the most promising assays which is increasingly accepted as a more sensitive indicator of myeloma disease status is the Minimal Residual Disease (MRD) analysis. Therefore, Investigators plan to use MRD analysis as a disease assessment tool throughout this study and will correlate it with conventional myeloma disease assessment tools. Investigators would also like to incorporate a newly developed assay - Heavy lite (HevyLite) Chain assay and to explore the feasibility of using optional cell free DNA (cfDNA) to detect and monitor response assessments in multiple myeloma, - which will be done at the same time points as the other disease assessments thereby allowing us to explore the viability of these assays in clinical practice.

INTERVENTIONS:

Conditioning Regimen IV Busulfan 3.2mg/kg or equivalent pharmacokinetics directed dose once daily as a 3-hour infusion on days -5, -4 and -3 (option 1) or on days -6, -5, -4 (option 2).IV Melphalan 140mg/m2 once on day -2 (for option 1) or day -3 ( for option 2) Maintenance Regimen Oral Lenalidomide 10 mg once daily for 28 days of a 28 days cycle for first three cycles and then dose escalation to 15 mg daily if clinically appropriate to do so.

STUDY ENDPOINTS

Primary:

• MRD negativity at day 100 post ASCT

Secondary:

* To determine the pattern of MRD analysis during lenalidomide maintenance.
* To determine the response rate using conventional immunoglobulin-based markers at day 100 post ASCT and best response using lenalidomide maintenance.
* To determine the effectiveness of using the Heavy lite (HevyLite) Chain assay to assess anti-tumour response at day 100 post ASCT and during lenalidomide maintenance.
* To determine the toxicity of busulfan and melphalan when used as a high-dose conditioning therapy for ASCT.
* To determine the toxicity of lenalidomide maintenance post busulfan and melphalan conditioning ASCT.
* To determine the progression free survival (PFS) and overall survival (OS) of this program.
* To determine, through whole exome sequencing in individual Multiple Myeloma (MM) patients, the type and frequencies of somatic abnormalities (point mutations, indels, and copy number abnormalities) and their evolution overtime as the clinical disease progresses.
* To explore the feasibility of using optional cell free DNA (cfDNA) to detect and monitor response assessments in multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years, inclusive.
2. Study participants must have a diagnosis of symptomatic multiple myeloma requiring systemic therapy and are eligible for the planned ASCT.
3. Untreated bone marrow sample was shipped to Princess Margaret Hospital for MRD assay.
4. Must have been treated with a velcade-based induction regimen. No limit to the number of cycles of induction.
5. Study participants in whom the minimum stem cell dose of 2.0 x 106 cluster of differentiation (CD)34+ cells/kg has been collected.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
7. Negative beta-human chorionic gonadotropin (β-HCG) pregnancy test in all females of child-bearing potential (FOCBP).
8. Ability to provide written informed consent prior to initiation of any study-related procedures, and ability, in the opinion of the Principal Investigator, to comply with all requirements of the study.

Exclusion Criteria:

1. Myeloma progression at any time since starting initial induction therapy for multiple myeloma. Changes to or additions to the existing induction therapy are allowed as long as disease progression has not been confirmed.
2. Prior treatment history of ASCT for any medical reason.
3. Prior treatment history of high-dose chemotherapy with stem cell rescue for any medical reason, not limited to myeloma treatment.
4. Prior treatment with busulfan or gemtuzumab ozogamicin for any reason.
5. Systemic amyloidosis.
6. Left ventricular ejection fraction (LVEF) < 45% as measured by either multi-gated acquisition scan (MUGA) or echocardiogram (ECHO) performed within 75 days prior to day of busulfan dose. If cyclophosphamide was used for stem cell harvest, an ECHO or MUGA must be done after the stem cell collection and prior to enrollment to confirm adequate cardiac function.
7. Uncontrolled arrhythmia or symptomatic cardiac disease at the time of screening.
8. Symptomatic pulmonary disease, based on Forced Expiratory Volume in 1 Second (FEV1), Forced Vital Capacity (FVC) or Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) < 50% of predicted (corrected for hemoglobin) measured within 75 days prior to day of busulfan dose.
9. Aspartate transaminase (AST)/alanine transaminase (ALT) ≥ 3 x the upper limit of normal (ULN).
10. History of elevated total serum bilirubin >2 mg/dL that had been caused by previous chemotherapy at any point, or total bilirubin > 2.0 mg/dL at the time of screening with the exception of Gilbert's disease.
11. Hepatic synthetic dysfunction evidenced by prolongation of the prothrombin time as International Normalized Ratio (INR) ≥ 2.0 at the time of screening.
12. Any previous history of fulminant liver failure, cirrhosis, alcoholic hepatitis, esophageal varices, hepatic encephalopathy, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, and symptomatic biliary disease.
13. Prior total body irradiation therapy, or radiation therapy directly applied to the liver.
14. Patients with a known history of hepatitis B or hepatitis C should be on appropriate anti-viral therapy. Even so, these cases must be discussed with the sponsor and approval obtained prior to screening.
15. Known history of or current HIV infection, or active hepatitis B or c infection or any uncontrolled active infection of any kind at the time busulfan administration.
16. Serum creatinine >177 umol/L at the time of screening.
17. Women who are pregnant or lactating.
18. Current or history of drug and/or alcohol abuse.
19. Use of other investigational therapies within 30 days of enrollment in this study. Use of investigational therapies, other than the ones given as part of this protocol therapy, is not allowed during the study participation.
20. Clinically significant abnormality in medical history or upon examination that might interfere with the outcomes of the study in the opinion of the investigator.
21. Any patient, who in the opinion of the investigator, should not participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
• Minimal Residual Disease (MRD) negativity at day 100 post ASCT | day 100 post ASCT
  The conventional immunological markers used to define myeloma disease status have also been a subject of debate recently with some reports suggesting that more accurate disease assessment tools are needed to better decide on management of this disease. One of the most promising assays which is increasingly accepted as a more sensitive indicator of myeloma disease status is the Minimal Residual Disease (MRD) analysis. Therefore, Investigators plan to use MRD analysis as a disease assessment tool throughout this study and will correlate it with conventional myeloma disease assessment tools. Investigators would also like to incorporate a newly developed assay - Heavy lite (HevyLite) Chain assay - which will be done at the same time points as the other disease assessments thereby allowing us to explore the viability of this assay in clinical practice.

SECONDARY OUTCOMES:
• To determine the pattern, positivity (in terms of percentages) or negativity of MRD analysis during lenalidomide maintenance. | After ASCT at day 100, during maintenance therapy every 3 months at month 6, 9 and 12 after ASCT; and thereafter every 6 months until disease progression and at discontinuation.
  The conventional immunological markers used to define myeloma disease status have also been a subject of debate recently with some reports suggesting that more accurate disease assessment tools are needed to better decide on management of this disease. One of the most promising assays which is increasingly accepted as a more sensitive indicator of myeloma disease status is the Minimal Residual Disease (MRD) analysis. Therefore, Investigators plan to use MRD negativity analysis as a disease assessment tool throughout this study and will correlate it with conventional myeloma disease assessment tools. Investigators would also like to incorporate a newly developed assay - Heavy lite (HevyLite) Chain assay - which will be done at the same time points as the other disease assessments thereby allowing us to explore the viability of this assay in clinical practice.
• To determine the response rate using conventional immunoglobulin and monoclonal protein-based markers at day 100 post ASCT and best response using lenalidomide maintenance. | After ASCT at day 100, during maintenance therapy every 3 months at month 6, 9 and 12 after ASCT; and thereafter every 6 months until disease progression and at discontinuation.
  The response rate (Complete Response, Very Good Partial Response, Partial Response, Minimal Response and Stable Disease) will be assessed by using the European Group for Blood and Marrow Transplantation modified response criteria,with conventional immunoglobulin and monoclonal protein-based markers at day 100 post ASCT and best response using lenalidomide maintenance.
• To determine the effectiveness of using the HevyLite Chain assay to assess anti-tumour response at day 100 post ASCT and during lenalidomide maintenance | After ASCT at day 100, during maintenance therapy every 3 months at month 6, 9 and 12 after ASCT; and thereafter every 6 months until disease progression and at discontinuation.
  Immunoglobulin (Ig) A kappa, Immunoglobulin (Ig)A lambda, Immunoglobulin (Ig) A kappa/Immunoglobulin (Ig) A lambda ratio; Immunoglobulin (Ig) G Kappa, Immunoglobulin (Ig) G Lambda,Immunoglobulin (Ig) G kappa/Immunoglobulin (Ig) G lambda ratio; Immunoglobulin (Ig) M Kappa, Immunoglobulin (Ig) M Lambda and Immunoglobulin (Ig) M kappa/Immunoglobulin (Ig) M lambda ratio will be measured. These results will be correlated to standard Free Lite Chain assays performed at the same time points listed above.
• To determine the toxicity of busulfan and melphalan when used as a high-dose conditioning therapy for ASCT. | During conditioning therapy for ASCT. For schema option 1 this will be assessed at days -6, -5, -4, -3 and -2 prior ASCT. For schema option 2 this will be assessed at days -7, -6, -5, -4 and -3 prior ASCT.
  Toxicity of busulfan and melphalan will be determined by tracking occurrence of adverse events, serious adverse events and immediately reportable events based on the definitions listed in the protocol section 18.1 The severity of the toxicity will be graded according to the NCI Common Toxicity Criteria for Adverse Effects(CTCAE) version 3.0
• To determine the toxicity of lenalidomide maintenance post busulfan and melphalan conditioning ASCT. | After day 100 post ASCT, during the maintenance therapy every 3 months at month 6, 9 and 12 after ASCT; and thereafter every 6 months until disease progression and at discontinuation.
  Toxicity of lenalidomide maintenance will be determined by tracking occurrence of adverse events, serious adverse events and immediately reportable events based on the definitions listed in the protocol section 18.1 The severity of the toxicity will be graded according to the NCI CTCAE version 3.0
• To determine the progression free survival (PFS) and overall survival (OS) of this program. | From randomization patients will be followed for PFS every 3 months for the first year after ASCT and then every 6 months until disease progression. After they will be followed every year for O/S until death.
  These endpoints will be analyzed as time to event variables, which is defined as the time from transplant to death for OS and the time from transplant to the first occurrence of death or disease progression for PFS. The event free probabilities for these endpoints will be estimated by the product limit Kaplan Meier method. Subjects without events will be censored at the last followup for OS and at the last disease evaluation for PFS.
• Identification of the type and frequencies of somatic abnormalities (point mutations, indels, and copy number abnormalities) and their evolution overtime. | After ASCT at day 100, during maint. therapy q 3 months at month 6 and 12 after ASCT; and thereafter every 6 months until disease progression and at discontinuation.
  Whole genome sequencing will be performed centrally at intervals described under the time frame.
• Assessment of using optional cell free DNA (cfDNA) in peripheral blood to monitor and correlate response assessments in multiple myeloma. | After ASCT at day 100, during maint. therapy q 3 months at month 6, 9 and 12 after ASCT; and thereafter every 6 months until disease progression and at discontinuation.
  cell free DNA (cfDNA) will be performed centrally at intervals described under the time frame AND only for study participants for whom genomics whole exome sequencing) samples have been collected.

CONTACTS AND LOCATIONS:
Overall Officials: Donna E Reece, MD, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (10):
- Canada (10):
  - Cross Cancer Institute 11560 University Ave, Edmonton, Alberta
  - Vancouver General Hospital, Centennial Pavilion, 6th Floor, Vancouver, British Columbia
  - Saint John Regional Hospital, 5DN Research Department, 400 University Ave, Saint John, New Brunswick
  - Queen Elizabeth II Health Sciences Centre., Halifax, Nova Scotia
  - London Regional Cancer Program 790 Commissioners Road East, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Hôpital Maisonneuve-Rosemont, 5415, boul. de l'Assomption, Montreal, Quebec
  - Royal Victoria Hospital, MUHC Glen Site, Cedars Cancer Centre, Montreal, Quebec
  - Saskatoon Cancer Centre 20 Campus Drive, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
Un-identified IPD, pertaining to Serious Adverse Events, will be submitted to the DSMB for review. DSMB letters will be provided to the participating sites.
  Un-identified IPD could also be shared with Sub-investigators conducting correlative studies for this trial; that will be Dr. Suzanne Trudel and Dr. Rodger Tiedemann.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Current Study Protocol Amendment # 4 (v. date February 13, 21018), ICF(s), interim CSR have been submitted to the DSMB since the activation of this trial. DSMB meetings occur every 6 months. DSMB letters are provided to participating sites every 6 months after the DSMB meetings have occurred.
  IPD for correlative studies is provided ad-hoc on individual request for data analysis (i.e. submission of abstracts to conferences).
Access Criteria: No additional information will be shared